CLINICAL TRIAL: NCT06037824
Title: Influence of Compressive Cryotherapy Compared to Conventional Cryotherapy on Articular, Trophic and Functional Recovery After Total Knee Arthroplasty: a Randomized Controlled Study
Brief Title: Compressive Cryotherapy Versus Conventional Cryotherapy After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Formation en Masso-Kinésithérapie Saint Michel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IFMK01
Record Dates: First submitted 2023-08-31; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Knee Arthropathy; Cryotherapy Effect
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group received classic rehabilitation* + compressive cryotherapy
  * classic rehabilitation include passive and active of mobilization of knee and patella, treat arthrogenic muscular inhibition, learn to lock the quadriceps, progressive muscular strengthening of the periarticular muscles of the knee, stretching of the quadriceps and the posterior muscular chain, proprioceptive exercises with bi- and unipodal balance, transfer of support and resumption of the walking pattern.
  Interventions: Other: cryotherapy
- Control Group (Active Comparator): This group received classic rehabilitation* + classic cryotherapy
  *classic rehabilitation include passive and active of mobilization of knee and patella, treat arthrogenic muscular inhibition, learn to lock the quadriceps, progressive muscular strengthening of the periarticular muscles of the knee, stretching of the quadriceps and the posterior muscular chain, proprioceptive exercises with bi- and unipodal balance, transfer of support and resumption of the walking pattern.
  Interventions: Other: cryotherapy

INTERVENTIONS:
Other: cryotherapy — cryotherapy was added to rehabilitation*. One group received compressive cryotherapy and the other conventional cold pack cryotherapy.
  * rehabilitation includes (="classic rehabilitation") passive and active of mobilization of knee and patella, treat arthrogenic muscular inhibition, learn to lock the quadriceps, progressive muscular strengthening of the periarticular muscles of the knee, stretching of the quadriceps and the posterior muscular chain, proprioceptive exercises with bi- and unipodal balance, transfer of support and resumption of the walking pattern.

SUMMARY:
In the postoperative period of a total knee arthroplasty, subjects present limitations of articular amplitudes, swelling, pain and functional limitations. Functional rehabilitation is unanimously recommended, including the use of cryotherapy. However, there is no consensus regarding the methods of application of cryotherapy. Thus the objective of the study is to compare 2 cryotherapy techniques associated with a classic rehabilitation on the improvement of mobility, swelling, pain and functional parameters. The 2 cryotherapies were a compressive cryotherapy and a so-called classic cryotherapy by cold pack.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* First-line Total Knee Arthroplasty on an indication of knee osteoarthritis diagnosed by radio-clinical examination
* Between D3 and D10 postoperatively
* Age < 90 years.

Exclusion Criteria:

* Intolerance to cryotherapy or compression,
* Occurrence of complications secondary to surgery,
* Withdrawal of consent,
* Non-compliance with the rehabilitation protocol (content and dosage of sessions).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
knee range of motion | Day 1-Day 8-Day 15-Day 21
  Measurement of passive flexion and active extension with a goniometer

SECONDARY OUTCOMES:
Knee perimetry | Day 1-Day 8-Day 15-Day 21
  A perimetry measurement with a tape measure was carried out
Swelling | Day 1-Day 8-Day 15-Day 21
  Swelling has been measured with the "fluctuation test": the examiner placed his thumb and fingers on either side of the lower part of the patella, while with his other hand, he positioned himself at the level of the upper part of the sub quadriceps fornix. The fingers of the cranial hand exerted light pressure to mobilize the fluid from the quadriceps fornix. The test was positive if the fingers or thumb were pushed back by the effusion.
Pain at rest and on exertion | Day 1-Day 8-Day 15-Day 21
  Pain assessment was based on the use of the Verbal Numerical Scale (NVS). The examiner asked the subject to quantify their pain on a scale ranging from 0 to 10 (0 corresponding to no pain and 10 to unbearable pain). Pain assessment was carried out at rest and during exercise during the rehabilitation sessions.
6min walking test | Day 1-Day 8-Day 15-Day 21
  The instructions were to cover the greatest distance possible for 6 minutes
KOOS score (Knee injury and Osteoarthritis Outcome Score) | Day 1-Day 8-Day 15-Day 21
  Only the 17 items of the questionnaire dealing with "quality of life" were considered in this study. Subjects had to complete the questions

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Porte Verte, Versailles, Yvelines, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quesnot A, Mouchel S, Salah SB, Baranes I, Martinez L, Billuart F. Randomized controlled trial of compressive cryotherapy versus standard cryotherapy after total knee arthroplasty: pain, swelling, range of motion and functional recovery. BMC Musculoskelet Disord. 2024 Feb 28;25(1):182. doi: 10.1186/s12891-024-07310-7. PMID 38419032